CLINICAL TRIAL: NCT02512185
Title: TOward Personalizing Care for Older Men With mCRPC - Understanding and Predicting Treatment Toxicities (the TOPCOP Study)
Brief Title: Towards Optimal Prescription of Chemotherapy in Prostate Cancer
Acronym: TOPCOP
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Prostate Cancer Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 15-9075
Record Dates: First submitted 2015-07-17; First posted 2015-07-30 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Chemotherapy; mCRPC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chemotherapy: Men starting first-line chemotherapy for mCRPC (typically Docetaxel and Prednisone)
- Abiraterone: Men with mCRPC starting Abiraterone
- Enzalutamide: Men with mCRPC starting Enzalutamide

SUMMARY:
This study will examine the impact of modern treatments for metastatic Castrate Resistant Prostate Cancer (mCRPC) on several relevant 'geriatric' domains such as daily function, objective physical function, and falls. Additionally, the investigators study whether frailty is associated with worse outcomes, and whether it is possible to predict the risk of severe chemotherapy toxicity in older men.

DETAILED DESCRIPTION:
Our primary aims are (a) to examine the impact of pre-treatment frailty on 'elder-relevant' outcomes including daily function, objective physical function, falls, quality of life (QOL), and early treatment discontinuation; (b) to determine whether the Hurria/Cancer and Aging Research Group (CARG) tool is able to predict severe (grade 3+) chemotherapy toxicity in men starting chemotherapy. Our secondary aim is to understand the impact of abiraterone and enzalutamide on 'elder-relevant' outcomes.

This is a prospective multicentre observational study. The investigators will enroll men age 65 or older with mCRPC who are starting (a) first-line chemotherapy; (b) abiraterone; or (c) enzalutamide. Assessments will occur prior to starting treatment and every 2 months thereafter until the end of treatment.

As treatment options become more complex in older men with mCRPC, understanding and predicting a wide range of treatment toxicities is important and will aid decision-making and management.

ELIGIBILITY:
Inclusion Criteria:

1. At least 65 years of age
2. Diagnosed with prostate cancer with evidence of clinical and/or radiographic evidence of progression despite adequate androgen deprivation therapy and achievement of castration (total testosterone level <1.7 nmol/L measured within 6 months of enrollment)
3. Among men starting either abiraterone or enzalutamide, no prior chemotherapy/abiraterone/enzalutamide. Among men starting first-line chemotherapy, commencing docetaxel but can have had either prior abiraterone or enzalutamide

Exclusion Criteria:

1. Unable to speak English fluently.
2. Severe neuropsychiatric abnormalities that prevent study participation.
3. Limited life expectancy (<3 months) as estimated by the primary oncologist.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men 65 and older starting first line chemotherapy, or Abiraterone, or Enzalutamide for mCRPC
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Daily function assessed by questionnaires | Participants will be followed for the duration of treatment up to 2 years
  Daily function
Objective physical function | Participants will be followed for the duration of treatment up to 2 years
  Will be assessed by 3 physical performance measures
Grade 3+ toxicity using Common Terminology Criteria for Adverse Events (CTC-AE) version 4.0 | Participants will be followed for the duration of treatment up to 2 years
  Toxicity
Number of falls provided by the participant | Participants will be followed for the duration of treatment up to 2 years
  Falls
Body fat percentage will be measured using a Tanita 300A analyzer | Participants will be followed for the duration of treatment up to 2 years
  Body composition analysis

SECONDARY OUTCOMES:
Quality of Life (QOL) | Participants will be followed for the duration of treatment up to 2 years
  FACT-G and FACT-P (specific for prostate cancer) questionnaires will be administered
The Montreal Cognitive Assessment (MoCA test) and Trail making tests A&B | Participants will be followed for the duration of treatment up to 2 years
  Cognition composite

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre -KGH, Kingston, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No